CLINICAL TRIAL: NCT04097106
Title: Synbiotic Supplement Effects on Gastrointestinal Symptoms and Gut Microbiota and Fecal Metabolomics
Brief Title: Synbiotic Dietary Supplement and Gut Microbiota
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Gail Cresci, Director Nutrition Research within Center for Human Nutrition, The Cleveland Clinic
Other Study IDs: IRB #19-601
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lean BMI (19-25)
  Interventions: Dietary Supplement: Synbiotic
- Obese BMI (30-35)
  Interventions: Dietary Supplement: Synbiotic

INTERVENTIONS:
Dietary Supplement: Synbiotic — Synbiotic dietary supplement in capsule form

SUMMARY:
To test the feasibility and safety of our designer synbiotic on gastrointestinal symptoms and gut microbiota and fecal metabolomics.

DETAILED DESCRIPTION:
This will be a double-blinded, randomized, placebo-controlled paired crossover pilot study in healthy controls aimed to evaluate gastrointestinal tolerance of a synbiotic dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-25 (lean) and BMI 30-35 (obese)
* Age 18-45 years old
* subjects must be willing to consume oral dietary supplement and placebo daily for a total of 56 days,
* willing to complete gastrointestinal (GI) and dietary surveys, body composition assessment, and provide blood, urine and stool sample at 4 intervals during the pilot study (baseline, after first supplementation period (day 28), after washout period (day 49), and after second supplementation period (day 77)

Exclusion Criteria:

* antibiotic consumption within 28 days of study initiation
* diabetes
* kidney disorders
* history of cardiac disease and medications for cardiac disease
* use of statins and antihypertensive drugs
* inflammatory bowel disease
* irritable bowel syndrome
* history of small intestinal bacterial overgrowth
* history of intestinal surgery, excluding hernia repair and appendectomy
* active cancer diagnosis; chronic acid suppression treatment (proton pump inhibitors, histamine H2 receptor antagonists)
* immune modulatory treatments (e.g. chronic immunosuppressive medications, chronic NSAIDs)
* abnormal liver or kidney function as measured by routine serum chemistry testing
* severe anemia or significant white blood cell or platelet abnormalities
* no additional blood or blood product donations during study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thirty two healthy volunteers, aged 18-45 years old, will be recruited for this pilot study, plan to enroll 16 subjects with a BMI 19-25 kg/m2 and 16 subjects with a BMI 30-35 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Measure change in gastrointestinal symptoms using "Rating of Gastrointestinal (GI) Symptoms" scale | Baseline, Day 28, day 49, day 77
  Rating of GI Symptoms scale includes 5 questions, which range from 0 (never affected) to 7 (always bothered), summed to compute total score
Change in microbiome stool diversity | Baseline, Day 28, day 49, day 77
Change in metabolome stool profile | Baseline, Day 28, day 49, day 77
Change in metabolome urine profile | Baseline, Day 28, day 49, day 77

CONTACTS AND LOCATIONS:
Overall Officials: Gail Cresci, Principal Investigator — The Cleveland Clinic
Locations (1):
- Kassandra Spates-Harden, Cleveland, Ohio, United States